CLINICAL TRIAL: NCT02148263
Title: Contact Lens Adaptation in Neophytes
Acronym: CLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Andrew Pucker, Senior Research Associate, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014H0074; K08EY023264 (NIH)
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Contact Lens Comfort
Keywords: Contact Lenses; Neophytes; Contact Lens Adaptation; Randomized

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full-Time Senofilcon A Contact Lens Wear (Experimental): This group will start wearing contact lenses 8 or more hours per day on the first day of wear
  Interventions: Device: senofilcon A
- Graduated Senofilcon A Contact Lens Wear (Experimental): This group will start wearing contact lenses on a graduated schedule (day 1 = 2 hours, day 2 = 4 hours, day 3 = 6 hours, day 4 = 8 hours, day 5 = 8 or more hours).
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A
  Other Names: Acuvue Oasys

SUMMARY:
Eye care professionals prescribe contact lenses to new wearers on a daily basis, and it is common practice for practitioners to educate their patients to gradually increase their contact lens wear time over their first few days of use; however, there is no scientific basis in the literature for this practice. This study will compare the ocular health and comfort of new contact lens wearers who are randomly assigned to begin contact lens wear with increasing wearing time versus those who immediately start full-time wear (eight hours or more/day). The increasing wearing time group will wear daily wear contact lenses (Acuvue Oasys) for two, four, six, eight, and eight or more hours on the first, second, third, fourth, and fifth days, respectively. The other group will be instructed to wear the same contact lenses for eight or more hours per day, starting with the first day of wear. Both groups of subjects will have their eye health and comfort evaluated at baseline, one, and two weeks with a lighted-microscope and eye comfort surveys. Subjects will also keep a daily log of eye comfort with a visual analog scale survey at home. All subjects will learn how to wear and take care of contact lenses. They will also receive a prescription for contact lenses at the conclusion if they wish to continue wearing the study contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Has had a completed comprehensive eye exam within the past 6 months
* Able to wear spherical senofilcon A contact lenses
* Able to use Opti-Free PureMoist contact lens solution

Exclusion Criteria:

* Any prior contact lens use
* Topical eye drops within the last two hours of the study visit
* Known systemic health conditions known to alter tear film physiology
* History of severe ocular trauma
* Active ocular infection
* Active ocular inflammation
* Known hypersensitivity to diagnostic eye drops
* Pregnant or breast feeding

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pucker, OD, MS, Principal Investigator — Ohio State University; Jeffrey J Walline, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Sullivan BD, Whitmer D, Nichols KK, Tomlinson A, Foulks GN, Geerling G, Pepose JS, Kosheleff V, Porreco A, Lemp MA. An objective approach to dry eye disease severity. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6125-30. doi: 10.1167/iovs.10-5390. Epub 2010 Jul 14. PMID 20631232
- [Background] Sullivan BD, Crews LA, Sonmez B, de la Paz MF, Comert E, Charoenrook V, de Araujo AL, Pepose JS, Berg MS, Kosheleff VP, Lemp MA. Clinical utility of objective tests for dry eye disease: variability over time and implications for clinical trials and disease management. Cornea. 2012 Sep;31(9):1000-8. doi: 10.1097/ICO.0b013e318242fd60. PMID 22475641
- [Background] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260
- [Background] Yang SN, Tai YC, Sheedy JE, Kinoshita B, Lampa M, Kern JR. Comparative effect of lens care solutions on blink rate, ocular discomfort and visual performance. Ophthalmic Physiol Opt. 2012 Sep;32(5):412-20. doi: 10.1111/j.1475-1313.2012.00922.x. Epub 2012 Jul 7. PMID 22775005
- [Background] Dougherty BE, Nichols JJ, Nichols KK. Rasch analysis of the Ocular Surface Disease Index (OSDI). Invest Ophthalmol Vis Sci. 2011 Nov 7;52(12):8630-5. doi: 10.1167/iovs.11-8027. PMID 21948646
- [Background] Chalmers RL, Begley CG. Dryness symptoms among an unselected clinical population with and without contact lens wear. Cont Lens Anterior Eye. 2006 Mar;29(1):25-30. doi: 10.1016/j.clae.2005.12.004. Epub 2006 Jan 31. PMID 16448840
- [Background] Faber E, Golding TR, Lowe R, Brennan NA. Effect of hydrogel lens wear on tear film stability. Optom Vis Sci. 1991 May;68(5):380-4. doi: 10.1097/00006324-199105000-00010. PMID 1852401
- [Background] Efron N, Morgan PB, Katsara SS. Validation of grading scales for contact lens complications. Ophthalmic Physiol Opt. 2001 Jan;21(1):17-29. PMID 11220037
- [Derived] Pucker AD, Steele K, Rueff E, Franklin QX, McClure K, Savla K, Walline JJ. Contact Lens Adaption in Neophytes. Optom Vis Sci. 2021 Mar 1;98(3):266-271. doi: 10.1097/OPX.0000000000001662. PMID 33771956

RESULTS

PARTICIPANT FLOW:
Groups:
- Full-Time Senofilcon A Contact Lens Wear: This group will start wearing contact lenses 8 or more hours per day on the first day of wear
  senofilcon A
- Graduated Senofilcon A Contact Lens Wear: This group will start wearing contact lenses on a graduated schedule (day 1 = 2 hours, day 2 = 4 hours, day 3 = 6 hours, day 4 = 8 hours, day 5 = 8 or more hours).
  senofilcon A
Period: Overall Study
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Started | 12 | 13
Completed | 9 | 11
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 22.8 [14 to 25] | 24.1 [20 to 29] | 23.45 [14 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 9 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Between-Group Difference in Eye Comfort as Measured by the Ocular Surface Disease Index (OSDI)
Description: This is an eye comfort survey. The Ocular Surface Disease Index (OSDI) is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
Units on a Scale | 10.8 (8.5) | 16.3 (18.8)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Between-Group Difference in Visual Acuity as Measured With the Bailey-Lovie Chart
Description: The investigator will measure the subject's visual acuity with a Bailey-Lovie high-contrast paper (logMAR) chart. logMAR is a method used to observe visual acuity. Smaller numbers are better scores.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
units on a scale | 0.03 (0.05) | 0.01 (0.08)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Between-Group Difference in Tear Stability as Measured by Non-Invasive Break Up Time (NIBUT)
Description: Non-Invasive Break Up Time (NIBUT) is a measure of tear stability. The range is 0 to 60 seconds with longer times being better tear stability.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
seconds | 11.7 (7.0) | 9.8 (2.7)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear; Test type: Superiority; p = .94, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Between-Group Difference in Tear Volume as Measured by Tear Meniscus Height (TMH)
Description: Tear Meniscus Height (TMH) was used at a measure of tear volume. The range is 0.0 to 2.0 mm with higher values being more tear volume.
Time Frame: 2 Weeks
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
mm | 0.31 (0.09) | 0.32 (0.12)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = .96, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Between-Group Difference in Bulbar Conjunctival Redness as Measured With the Keratograph 5M
Description: Eye redness was measured via bulbar conjunctival redness as measured with the Keratograph 5M. The range is 0 to 4 units with lower numbers being better.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
units on a scale | 0.69 (0.37) | 0.59 (0.09)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = .14, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Between-Group Difference in Upper and Lower Eyelid Blepharitis
Description: A slit-lamp biomicroscope was used to document eyelid blepharitis with a 0-3 scale by each eyelid with higher scores being worse blepharitis.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
units on a scale
  Two Weeks (Upper Eyelid) | 1.1 (1.3) | 1.3 (0.8)
  Two Weeks (Lower Eyelid) | 0.4 (0.7) | 0.8 (0.8)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority — This is for the upper eyelid evaluation; p = .27, Fisher Exact
Statistical Analysis 2: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; This is for the lower eyelid evaluation; Test type: Superiority; p = .58, Fisher Exact

7. Secondary Outcome: Between-Group Difference in Corneal Sodium Fluorescein Staining
Description: The Brien Holden Vision Institute grading scale was used to evaluate staining by observing the eye after applying sodium fluorescein. Scores were given for the extent (0-20 units), depth (0-20 units), type (0-20 units) of staining. Higher scores indicate worse staining.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
units on a scale
  Two Weeks (Extent) | 0.0 (0.1) | 0.3 (0.4)
  Two Weeks (Type) | 0.0 (0.0) | 0.2 (0.4)
  Two Weeks (Depth) | 0.0 (0.1) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Extent; Test type: Superiority; p = .50, Fisher Exact
Statistical Analysis 2: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Type; Test type: Superiority; p = .76, Fisher Exact
Statistical Analysis 3: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Depth; Test type: Superiority; p = .50, Fisher Exact

8. Secondary Outcome: Between-Group Difference in Tear Volume as Measured by Schirmer's Test I
Description: Tear volume was assessed with Schirmer's Test I test over 5 mins. This test has a 0-35 mm range with higher values being better tear volume.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
mm | 15.9 (8.8) | 21.2 (12.5)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Between-Group Difference in End of Day Contact Lens Comfort as Measured With a Visual Analog Scale (VAS)
Description: End of day contact lens comfort was measured with a visual analog scale (1-100 scale). Higher scores indicate better comfort.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 9 | 11
score on a scale | 89.0 (9.7) | 81.8 (18.7)
Statistical Analysis 1: Comparison: Full-Time Senofilcon A Contact Lens Wear vs Graduated Senofilcon A Contact Lens Wear; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Between-Group Difference in Contact Lens Dry Eye-8 Questionnaire (CLDEQ-8) Scores
Description: Contact lens comfort was measured with a scale (1-37 scale). Lower scores indicate better comfort.
Time Frame: 2-Weeks
Population: The electronic data capture system did not record these data correctly, so we could not analyze it. Therefore, data from the CLDEQ-8 are not valid.
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Full-Time Senofilcon A Contact Lens Wear | Graduated Senofilcon A Contact Lens Wear
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
There was a data collection error, which prevented the study from analyzing CLDEQ-8 scores. This study also intended to included conjunctival staining with lissamine green; however, lissamine green was not available during the conduct of this study, so this outcome was not included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02148263/Prot_SAP_ICF_000.pdf